CLINICAL TRIAL: NCT06978621
Title: Immunogenicity and Safety of Inactivated Hepatitis A Vaccine in Healthy Thai Children and Adolescents Lacking Protective Antibody Levels After a Single Dose of Live-attenuated Hepatitis A Vaccine
Brief Title: Immunogenicity and Safety of I-HAV in Healthy Thai Children and Adolescents Lacking Protective Antibody After L-HAV
Acronym: HAV-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Collaborators: Faculty of Medicine, Chiang Mai University (Unknown)
Responsible Party: Principal Investigator, Tavitiya Sudjaritruk, Associate Professor, Chiang Mai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PED-2568-0180
Record Dates: First submitted 2025-04-30; First posted 2025-05-18 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Hepatitis A; Hepatitis A Virus; Vaccine-Preventable Diseases
Keywords: Inacitivated hepatitis A vaccine; Safety; Immunogenicity; Clinical trial
MeSH Terms: conditions — Hepatitis A; Hepatitis; Vaccine-Preventable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inactivated HAV vaccine (I-HAV) (Experimental): An additional dose of inactivated hepatitis A vaccination for participants who have seronegative (anti-HAV IgG <1 S/CO) at baseline (1 year after a single dose of live-attenuated hepatitis A vaccine).
  Interventions: Biological: Inactivated hepatitis A vaccine (I-HAV)

INTERVENTIONS:
Biological: Inactivated hepatitis A vaccine (I-HAV) — A formaldehyde-inactivated hepatitis A virus (HM175 hepatitis A virus strain)
  Dose and administration: 0.5 mL intramuscular injection for participants age <=18 years, and 1.0 mL intramuscular injection for participants age 19 years and above.

SUMMARY:
Hepatitis A virus (HAV) remains a common infection in Thai children. Two HAV vaccines are available: inactivated vaccine (I-HAV, 2 doses) and live-attenuated vaccine (L-HAV, single dose), but neither is included in Thailand's national immunization program. Our previous randomized, active-controlled, open-label, non-inferiority trial trial found that some participants remained seronegative after one L-HAV dose (anti-HAV IgG <1 S/CO) (preliminary data). This study aims to evaluate the immunogenicity and safety of an additional dose of I-HAV in healthy Thai children and adolescents who did not develop protective antibody levels after a single dose of L-HAV.

DETAILED DESCRIPTION:
Hepatitis A virus (HAV) infection remains a common cause of viral hepatitis among children and adolescents in developing countries, including Thailand. Currently, two types of HAV vaccines are available in Thailand; (1) inactivated HAV vaccine (I-HAV) which is recommended as a 2-dose series administered 6 months apart, approved for use in children aged 1 year and older, and (2) live-attenuated HAV vaccine (L-HAV) which is recommended as a single dose, approved for children aged 18 months and older. However, as neither vaccine is included in Thailand's Expanded Programme on Immunization (EPI), the national vaccination coverage remains suboptimal.

In 2024, the investigators conducted a randomized, active-controlled, open-label, non-inferiority trial to compare the immunogenicity and safety of the currently marketed I-HAV and L-HAV in healthy Thai children and adolescents aged 18 months to 18 years. Preliminary results showed that a proportion of participants remained seronegative following a single dose of L-HAV (anti-HAV IgG <1 S/CO). Based on these findings, the investigators hypothesize that an additional dose of I-HAV may be necessary to achieve adequate seroprotection in this population. Therefore, the aim of this study is to evaluate the immunogenicity and safety of an additional dose of I-HAV in healthy Thai children and adolescents who did not develop protective antibody levels after a single dose of L-HAV.

ELIGIBILITY:
Inclusion Criteria:

* Thai children and adolescents who previously participated in the previous RCT study
* Previously randomized to receive one dose of L-HAV vaccine within the past 1 year (+/- 2 months)
* Have not demonstrate a seropositivity against HAV (anti-HAV IgG <1 S/CO) at 1 month after L-HAV vaccination
* Participants and/or caregivers gives written inform consent/assent form

Exclusion Criteria:

* History of acute illness within 4 weeks prior to study enrollment
* Has a history of illness or a diagnosis consistent with hepatitis A after receiving the live attenuated hepatitis A vaccine as part of participation in a previous research study
* Has a history of receiving any additional hepatitis A vaccine after participating in the previous research study
* Presence of fever (body temperature ≥38.0°C), jaundice, or yellowing of the eyes within 4 weeks prior to study enrollment
* Has underlying conditions including thrombocytopenia, coagulopathy, hemophilia A or B, neurological disorders, immunodeficiency disorders, chronic liver disease, or chronic hepatitis B or C infection
* Has received immunosuppressive agents, immunomodulatory agents, or high-dose corticosteroids (greater than 2 mg/kg/day or more than 20 mg/day) for more than 14 consecutive days within 6 months prior to study enrollment
* Has received blood products or blood components, including immunoglobulins, within 6 months prior to study enrollment
* Has received other live vaccines within 30 days prior to study enrollment
* Has history of allergy to vaccines or any vaccine components, such as aluminum hydroxide, 2-phenoxyethanol, neomycin, formaldehyde, or gentamicin sulfate, or has history of severe allergic reactions (e.g., anaphylaxis) to any vaccines
* Women planning for pregnancy, pregnant women or lactating women
* Women in childbearing age who cannot use contraceptive methods during study participation
* Is concurrently involved in other clinical trials in which receiving an investigational vaccine or study drug as part of study participation
* Have any condition that, in the opinion of the site investigator, would compromise the subject's ability to participate in the study

Ages: 18 Months to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05-25 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Anti-HAV immunoglobulin G (IgG) seropositivity rate | at baseline (1 year after L-HAV vaccination) and 4 weeks after an additional I-HAV vaccination.
  Anti-HAV IgG seropositivity rate (anti-HAV IgG >= 1.0 S/CO) before and after an additional dose of I-HAV vaccine.
Incidence of adverse events following I-HAV vaccination | immediate and until 4 weeks after an additional I-HAV vaccination.
  Adverse events, including solicited local and systemic reactions as well as serious adverse events, following an additional dose of I-HAV vaccine.

SECONDARY OUTCOMES:
Geometric mean concentration (GMC) of anti-HAV IgG level | at baseline (1 year after L-HAV vaccination) and 4 weeks after an additional I-HAV vaccination.
  Geometric mean concentration (GMC) of anti-HAV IgG level before and after an additional dose of I-HAV vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Tavitiya Sudjaritruk, MD, PhD, Study Chair — Department of Pediatrics, Faculty of Medicine, Chiang Mai University; Natchaya Kunanitthaworn, MD, Principal Investigator — Department of Pediatrics, Faculty of Medicine, Chiang Mai University
Locations (1):
- Department of Pediatrics, Faculty of Medicine, Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available to other researchers for this study.

REFERENCES:
- [Background] Kunanitthaworn N, Mueangmo O, Saheng J, Wongjak W, Lertsiriladakul T, Chaito T, Nantarat P, Sudjaritruk T. Seroprevalence of hepatitis A virus antibodies among children and adolescents living in Northern Thailand: an implication for hepatitis A immunization. Sci Rep. 2023 Oct 13;13(1):17432. doi: 10.1038/s41598-023-44643-0. PMID 37833325
- [Background] Ma F, Yang J, Kang G, Sun Q, Lu P, Zhao Y, Wang Z, Luo J, Wang Z. Comparison of the safety and immunogenicity of live attenuated and inactivated hepatitis A vaccine in healthy Chinese children aged 18 months to 16 years: results from a randomized, parallel controlled, phase IV study. Clin Microbiol Infect. 2016 Sep;22(9):811.e9-811.e15. doi: 10.1016/j.cmi.2016.06.004. Epub 2016 Jun 23. PMID 27345175
- [Background] Liu XE, Wushouer F, Gou A, Kuerban M, Li X, Sun Y, Zhang J, Liu Y, Li J, Zhuang H. Comparison of immunogenicity between inactivated and live attenuated hepatitis A vaccines: a single-blind, randomized, parallel-group clinical trial among children in Xinjiang Uighur Autonomous Region, China. Hum Vaccin Immunother. 2013 Jul;9(7):1460-5. doi: 10.4161/hv.24366. Epub 2013 Apr 9. PMID 23571173